CLINICAL TRIAL: NCT02790190
Title: Phase III Study of Individualized Adaptive Radiotherapy Based on PET/CT and 3DCRT/IMRT in Combination With Chemotherapy for Locally Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Individualized Adaptive Radiotherapy Based on PET/CT and IMRT for Locally Advanced Non-Small Cell Lung Cancer (NSCLC)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Jinming Yu, president, Shandong Cancer Hospital and Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRTOG1601
Record Dates: First submitted 2016-05-29; First posted 2016-06-03 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-05

CONDITIONS: Lung Neoplasms
MeSH Terms: conditions — Lung Neoplasms

ARMS (2):
- Individualized Adaptive radiotherapy (Experimental): GTV dose per fraction will be 2.2-2.4 y per fraction for 20 fractions and PTV dose per fraction will be 2.0 Gy per fraction.Perform PET/CT before radiotherapy and at 36 Gy for treatment response assessment and adaptive plan.Adaptive plan treated at 2.2-3.8 Gy per fraction for GTV and 2.0 Gy for PTV in the final 10 fractions.
  Interventions: Other: Radiotherapy dose
- Conventional radiotherapy (No Intervention): 2 Gy per fraction for all patient,perform PET/CT before radiotherapy and at 40 Gy for treatment response assessment .Continue treatment to a total dose of 60 Gy.

INTERVENTIONS:
Other: Radiotherapy dose
  Arms: Individualized Adaptive radiotherapy

SUMMARY:
This is a perspective, multicenter,randomized controlled trial to compare the efficacy and safety of radiotherapy Based on PET/CT and IMRT combined with concurrent chemotherapy in patients with locally advanced non small cell lung cancer . Analyses of overall survival (OS) will be done as defined in the protocol.

DETAILED DESCRIPTION:
https://register.clinicaltrials.gov/prs/app/template/Home.vm?uid=U000184Z&ts=76&sid=S0006AP2&cx=r0ratc

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically proven non-small cell lung cancer.
2. Patients must be clinical AJCC stage IIIA or IIIB (AJCC, 7th ed.) with non-operable disease; non-operable disease will be determined by a multidisciplinary treatment team.
3. Patients with multiple, ipsilateral pulmonary nodules (T3, or T4) are eligible if a definitive course of daily fractionated RT is planned.
4. Appropriate stage for protocol entry, including no distant metastases, based upon the following minimum diagnostic workup:

   1. History/physical examination, including documentation of weight, within 2 weeks prior to registration;
   2. CT scan or sim CT of chest and upper abdomen (IV contrast is recommended unless medically contraindicated) within 6 weeks prior to registration;
   3. CT scan of the brain (contrast is recommended unless medically contraindicated) or MRI of the brain within 6 weeks prior to registration;
   4. Pulmonary function tests, including DLCO, within 6 weeks prior to registration; patients must have FEV1 ≥ 1.2 Liter or ≥ 50% predicted without bronchodilator;
   5. Zubrod Performance Status 0-1 within 2 weeks prior to registration;
   6. Age ≥ 18;
   7. Able to tolerate PET/CT imaging required to be performed at an ACR Imaging Core Lab qualified facility;
   8. CBC/differential obtained within 2 weeks prior to registration on study, with adequate bone marrow function;
5. Serum creatinine within normal institutional limits or a creatinine clearance ≥ 60 ml/min within 2 weeks prior to registration;
6. The patient must provide study-specific informed consent prior to study entry.

Exclusion Criteria

1. Any component of small cell lung carcinoma.
2. Evidence of a malignant pleural or pericardial effusion .
3. Prior invasive malignancy (except nonmelanomatous skin cancer) in 3 years ;
4. Prior systemic chemotherapy for the study cancer; note that prior chemotherapy for a different cancer is allowable.
5. Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields;
6. Severe, active co-morbidity, defined as follows:

   Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months; Transmural myocardial infarction within the last 6 months; Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration; Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; note, however, that laboratory tests for liver function and coagulation parameters are not required for entry into this protocol; Acquired Immune Deficiency Syndrome (AIDS) based upon current CDC definition; note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive. Protocol-specific requirements may also exclude immuno-compromised patients.
7. Pregnancy or women of childbearing potential and men who are sexually active and not willing to use medically acceptable forms of contraception.
8. Poorly controlled diabetes (defined as fasting glucose level > 200 mg/dL) ;
9. Patients with T4 disease with radiographic evidence of massive invasion of a large pulmonary artery and tumor causing significant narrowing and destruction of that artery are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 24 months

SECONDARY OUTCOMES:
Progression free survival | 24 months
Objective response rate | 24 months
local control rate | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Shuanghu Yuan, Ph.D ， M.D, Study Director — Shandong Cancer Hospital and Institute
Locations (24):
- China (24):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Fujian Province Cancer Hospital, Fuzhou, Fujian
  - the First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Liuzhou worker's hospital, Liuchow, Guangxi
  - Fourth hospital of hebei medical university, Shijiazhuang, Hebei
  - the second Hospital of hebei medical University, Shijiazhuang, Hebei
  - The Affiliated tumour Hospital of haerbin Medical University, Haerbin, Heilongjiang
  - The Affiliated Cancer Hospital of Zhengzhou University, Zhengzhou, Henan
  - Wuhan Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Hubei Provincial Renmin Hospital, Wuhan, Hubei
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Qianfoshan Hospital of Shandong, Jinan, Shandong
  - Shandong Cancer Hospital and Institute, Jinan, Shandong
  - The affiliated hospital of qingdao university, Qingdao, Shandong
  - Teng Zhou Central People's Hospital, Tengzhou, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Xijing hopital, Xi’an, Shanxi
  - the Affiliated Hospital of southwest medicalUniversity, Luzhou, Sichuan
  - The Affiliated Tumor Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The First People's Hospital of Hangzhou, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Medical School of Zhejiang University, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - the First Affiliated Hospital of wenzhou medical University, Wenzhou, Zhejiang